CLINICAL TRIAL: NCT04702347
Title: Genetic Testing in Upper Tract Urothelial Carcinoma (UTUC): the Epicheck Study
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Fundacio Puigvert (Other)
Collaborators: Nucleix Ltd. (Industry)
Responsible Party: Principal Investigator, Alberto Breda, Chief of the Uro-Oncology Unit and Director of the Kidney Transplantation Division, Fundacio Puigvert
Other Study IDs: C2018/35
Record Dates: First submitted 2021-01-04; First posted 2021-01-08 (Actual); Last update posted 2021-01-08 (Actual); Status verified 2021-01

CONDITIONS: Urologic Cancer; Urologic Neoplasms
Keywords: Upper tract urothelial carcinoma; Urinary biomarker; Liquid biopsy; Epigenetics; Surveillance; Follow-up
MeSH Terms: conditions — Urologic Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Urine from upper urinary tract and bladder (at least 10 ml each)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: Urine biomarker — Bladder urine samples (> 10 ml) will be collected for cytology and for the methylation test before cystoscopy. Prior to semirigid and flexible ureteroscopy, urine specimens from the upper urinary tract will be obtained via a ureteral catheter.

SUMMARY:
Background:

Upper tract urothelial carcinoma (UTUC) is a rare tumor associated with bladder cancer in up to 50% of cases. Its incidence is rising due to improved detection and bladder cancer survival. The diagnosis of UTUC is challenging because more than 35% of the standard biopsies can result inconclusive. The grading of UTUC cells, which delivers the most important data for the choice between a kidney-sparing surgery (KSS) and a radical treatment, is upgraded in 30% of radical nephroureterectomies. The follow-up of UTUC after KSS requires an invasive procedure as a diagnostic ureteroscopy for a minimum of 5 years, and urinary cytology has low diagnostic power.

Objective:

The aim of the study is to evaluate the accuracy (overall and stratified for grade) of a DNA methylation urine biomarker test (Bladder EpiCheckTM) in UTUC, and to compare it with current standard (urinary cytology). The secondary objective is to show its applicability in the specific clinical scenario of UTUC surveillance after kidney-sparing surgery and related cost-effectiveness.

Design, Setting, and Participants:

From February 2019 to February 2021, 80 consecutive patients candidates to ureteroscopy for suspicion of primary, recurrent or metachronous UTUC in one tertiary Referral Centers (Fundaciò Puigvert) giving written informed consent will be included in the study.

Intervention:

Bladder urine samples (> 10 ml) will be collected for cytology and for the methylation test before cystoscopy. Prior to semirigid and flexible ureteroscopy, urine specimens from the upper urinary tract will be obtained via a ureteral catheter.

ELIGIBILITY:
Inclusion Criteria:

* Patients suspected for primary or recurrent upper tract urothelial cancer requiring ureteroscopy

Exclusion Criteria:

* Metastatic disease with patient unfit for ureteroscopy
* Positive cystoscopy (concomitant presence of bladder cancer)
* Macroscopic hematuria not self-limiting requiring upfront nephroureterectomy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patients candidate to ureteroscopy for a radiological diagnosis or clinical suspicion for upper tract urothelial cancer in the period from February 1st 2019 to February 28th 2021 will be included in this study after giving informed written consent.
Sampling Method: Probability Sample
Enrollment: 80 (Estimated)
Dates: Start 2019-02-01 (Actual); Primary Completion 2021-02-28 (Estimated); Study Completion 2021-02-28 (Estimated)

PRIMARY OUTCOMES:
Sensitivity, specificity, positive predictive value and negative predictive value of the test | Through study completion, an average of 1 year
  To test the accuracy of the urine biomarker
Comparison with urinary cytology | Through study completion, an average of 1 year
  To evaluate and compare performance of urinary cytology and urine biormarker
Evaluation of biormarker performance in bladder and upper tract | Through study completion, an average of 1 year
  To compare the accuracy of the test in situ (upper tract) and in the bladder

SECONDARY OUTCOMES:
High grade/low grade tumors diagnosis | Through study completion, an average of 1 year
  Sub-analysis on biormaker accuracy for low and high grade tumours
Impact of the urine biormaker for UTUC diagnosis | Through study completion, an average of 1 year
  A decision-making analysis will be performed in patients with UTUC suspicion, reporting the net benefit, the number of unnecessary ureteroscopies avoided

CONTACTS AND LOCATIONS:
Locations (1):
- Fundacio Puigvert, Barcelona, Spain